CLINICAL TRIAL: NCT06199349
Title: Phase Ib Clinical Study on the Safety, Tolerability and Pharmacokinetic Characteristics of GMDTC for Injection After Repeated Administration in People With Excessive Cadmium Levels
Brief Title: Safety Study of GMDTC Injection in Participants With Excessive Cadmium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jianersheng (Zhuhai) Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: JianerShengPharmaTCIb
Record Dates: First submitted 2023-12-29; First posted 2024-01-10 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cadmium Exceeds the Standard
Keywords: cadmium; Cadmium Poisoning; Therapeutics; Drugs, Investigational; GMDTC
MeSH Terms: conditions — Cadmium Poisoning | interventions — Injections; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This clinical study is a double-blind study, in which participants such as clinical researchers, project managers, and project monitors are unaware of the random coding and drug administration groups of the subjects. Non-blind monitoring during the clinical study will be conducted by non-blind monitors. In addition, drug preparation will be carried out by non-blind researchers independent of this study. Analysis and testing personnel will also adopt blind analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GMDTC group (Experimental): The subjects assigned to the GMDTC group will be administered once every morning after eating a standard breakfast on D1-D3 and D8-D10.
  Interventions: Drug: GMDTC for injection
- Normal saline group (Placebo Comparator): The subjects assigned to the placebo group will be administered once every morning after eating a standard breakfast on D1-D3 and D8-D10.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: GMDTC for injection — GMDTC for injection with a specification of 0.5g/vial, 500mg,1000mg,2000mg, and administered by intravenous infusion. Using 0.9% physiological saline (0.5g will be prepared with 250mL injection solution to achieve a concentration of 2mg/mL). Using an infusion pump at a rate of 4mL/min according to the dosage, and any infusion reactions will be recorded. The injection solution for both the experimental and placebo groups should be prepared by a non-blind investigator independent of the trial.
  Other Names: GMDTC Group
  Arms: GMDTC group
Other: Normal saline — 0.9% physiological saline for injection with a specification of 250ml/bag, and administered by intravenous infusion. Using an infusion pump at a rate of 4mL/min according to the dosage, and any infusion reactions will be recorded. The injection solution for both the experimental and placebo groups should be prepared by a non-blind investigator independent of the trial
  Other Names: Normal saline group
  Arms: Normal saline group

SUMMARY:
This trial is a randomized, double-blind, single-center, single-dose escalating Phase I clinical trial designed to evaluate the safety, tolerability, and pharmacokinetic characteristics of GMDTC for injection after repeated administration in people with excessive cadmium levels.

DETAILED DESCRIPTION:
The primary objective of this study isto evaluate the safety and tolerability of injectable GMDTC for repeated administration in people with excessive cadmium. The secondary objective is to evaluate the pharmacokinetic and pharmacodynamic characteristics of GMDTC for injection in people with excessive cadmium levels after multiple administrations, and to explore the most effective dose. Based on the results of the single-dose study, three dose groups were designed, including a low-dose group, a medium-dose group, and a high-dose group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, both male and female are eligible;
* Male subjects must weigh at least 50.0 kg and female subjects must weigh at least 45.0 kg, with a body mass index (BMI) between 19 and 26 kg/m2, including the critical value;
* Urinary cadmium >5 μmol/mol creatinine for 2 consecutive days during the screening period (creatinine content is ≥0.3 μg/L and ≤3 μg/L).
* Subjects must voluntarily sign a written informed consent form.

Exclusion Criteria:

* Those who are currently suffering from any clinically serious disease and the researcher determines that there are safety risks in participating in this clinical trial;
* Those with eGFR<30 mL/min/1.73 m2 during screening (eGFR calculated using the Cockcroft-Gault formula: eGFR (mL/min/1.73 m2) =*(140-age) *weight (kg)/ [0.818*Cr (umol/L)] *0.85 (female));
* Those who have a history of allergies to 3 or more substances, or are allergic to any ingredients in this product；
* Those who have undergone surgical procedures within 4 weeks before screening or plan to undergo surgical procedures that affect pharmacokinetics and safety determination during the study period；
* Those who have taken any drugs or health care products that may interact with the experimental drugs within 14 days before screening (such as SGLT2 inhibitors such as dapagliflozin, canagliflozin, empagliflozin, empagliflozin, canagliflozin, etc.) Gliflozin, Henggliflozin, Ipagliflozin, Rupagliflozin, Togliflozin, and the natural compound phlorizin, etc.; GLUT2 inhibitors such as cytochalasin B, phloretin, Huoxiang Zhengqi Powder, and Mignonette herbalin and isoorientin, etc.);
* Those who have used any clinical trial drugs or enrolled in any drug/medical device clinical trials within 3 months before screening;
* Those who donated blood or suffered massive blood loss (≥200 mL, excluding female menstrual blood loss), received blood transfusions or used blood products within 3 months before screening;
* inability to tolerate venipuncture and/or history of fainting or needle phobia;
* pregnant or lactating women, and subjects who cannot adopt effective non-drug contraceptive measures during the study period;
* unable to adopt contraceptive measures within 6 months after the end of the study;
* have special dietary requirements and cannot adhere to a uniform diet;
* Alcoholics or regular drinkers within 6 months before screening, that is, drinking more than 14 units of alcohol per week (1 unit ≈ 200 mL of beer with an alcohol content of 5% or 25 mL of spirits with an alcohol content of 40%- or 85-mL wine with an alcohol content of 12%) or who cannot stop using any alcohol-containing products during the trial;
* unable to stop using any tobacco products during the study period;
* alcoholics or frequent drinkers within 6 months before screening, i.e., drinking more than 14 units of alcohol per week (1 unit - 360.5 mL of beer or 45 mL of 40% alcohol or 150 mL of wine) or unable to stop using any alcohol-containing products during the study period;
* drug abusers or those who used soft drugs (such as marijuana) within 3 months before screening or used hard drugs (such as cocaine, benzoyl peroxide, etc.) within 1 year before screening;
* Laboratory tests must meet one or more of the following during screening: white blood cell count<3.0×109/L, neutrophil count <1.5×109/L, red blood cell count <3.0×1012/L, hemoglobin<100 g/L , platelet count <1 × LLN, total bilirubin > 2 × ULN, alanine aminotransferase > 2 × ULN, aspartate aminotransferase >2 × ULN；
* The subjects may not be able to complete the study due to other reasons or the researchers believe that they should not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Adverse events | Up to 30 days
  Adverse events will be evaluated according to the NCI Common Terminology Criteria for Adverse Events (CTCAE, V5.0), which includes spontaneously reported adverse events as well as clinically significant changes in vital signs, physical examination, laboratory tests, electrocardiogram, and other examinations conducted during the trial.

SECONDARY OUTCOMES:
Pharmacokinetic parameters,Tmax | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  Peak time, reflecting the absorption, distribution, metabolism and excretion characteristics of drugs in the body.
Pharmacokinetic parameters, Cmax | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  Peak concentrations, reflecting the absorption, distribution, metabolism and excretion characteristics of drugs in the body.
Pharmacokinetic parameters, λz | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  The apparent terminal elimination rate constant, obtained by taking a half-log linear regression at the elimination phase concentration point, reflecting the absorption, distribution, metabolism and excretion characteristics of drugs in the body.
Pharmacokinetic parameters, t1/2 | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  the apparent terminal elimination half-life, calculated according to the following equation:t1/2= Ln(2)/ λz,reflecting the absorption, distribution, metabolism and excretion characteristics of drugs in the body.
Pharmacodynamic parameters, blood cadmium | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  blood cadmium concentration before and after drug administration
Pharmacodynamic parameters, urine cadmium | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  urine cadmium level before and after drug administration (μmol/mol creatinine)
Pharmacodynamic parameters, 24-hour urine cadmium | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  24-hour urine cadmium excretion before and after drug administration
Pharmacodynamic parameters,serum electrolyte and trace element | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  serum electrolyte and trace element concentrations before and after drug administration
Pharmacodynamic parameters, other blood heavy metals | Evaluated at baseline, during drug infusion, and within 24 hours after drug administration
  whole blood heavy metal levels before and after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Yan Lai, Principal Investigator — Hunan Occupational Disease Prevention and Control Institute; Fang Pei, PhD-c, Principal Investigator — Hunan Occupational Disease Prevention and Control Institute
Locations (1):
- Hunan Occupational Disease Prevention and Control Institute, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang X, Zhu J, Zhong Z, Luo M, Li G, Gong Z, Zhang C, Fei F, Ruan X, Zhou J, Liu G, Li G, Olson J, Ren X. Mobilization and removing of cadmium from kidney by GMDTC utilizing renal glucose reabsorption pathway. Toxicol Appl Pharmacol. 2016 Aug 15;305:143-152. doi: 10.1016/j.taap.2016.06.001. Epub 2016 Jun 6. PMID 27282297
- [Background] Li Guangxian. Study on the efficacy of GMDTC in removing cadmium and its toxic side effects in chronic cadmium-poisoned mice and rats [D]. Guangdong Pharmaceutical University, 2015.
- [Background] Guidelines for the management of Phase I clinical trials of drugs (trial implementation)